CLINICAL TRIAL: NCT00689962
Title: A Randomized, Prospective Comparison of Stainless Steel and Bioabsorbable Screw Fixation of Lisfranc Foot Injuries
Brief Title: A Comparison of Steel and Bioabsorbable Screw Fixation of Lisfranc Foot Injuries
Acronym: Lisfranc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Principal Investigator, Jamal Ahmad, Assistant Professor of Orthopaedic Surgery, Rothman Institute Orthopaedics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lisfranc 1
Record Dates: First submitted 2008-05-31; First posted 2008-06-04 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Joint Instability
Keywords: Lisfranc; fracture; dislocation; bioabsorbable
MeSH Terms: conditions — Joint Instability; Fractures, Bone; Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients with unstable Lisfranc foot fracture-dislocations that receive bioabsorbable screw fixation through surgery.
  Interventions: Device: Linvatec 4.5 mm Smart Screw
- 2 (Active Comparator): Patients with unstable Lisfranc fracture-dislocations of the foot that receive steel screw fixation through surgery.
  Interventions: Device: Synthes 4.0 mm steel screw

INTERVENTIONS:
Device: Linvatec 4.5 mm Smart Screw — Linvatec 4.5 mm Smart Screw to surgically fix the foot's Lisfranc ligaments
  Arms: 1
Device: Synthes 4.0 mm steel screw — Standard steel screw use to surgically fix the foot's Lisfranc ligaments.
  Arms: 2

SUMMARY:
I hypothesize that absorbable screw fixation of the foot's Lisfranc ligaments does not yield significant differences in postoperative foot stability, ligament function, and symptoms when compared to steel screw fixation. In addition, absorbable screw fixation of the Lisfranc ligaments offers the advantage that a second surgical procedure to remove the screw is not necessary.

DETAILED DESCRIPTION:
The Lisfranc ligaments are a group of ligaments that connect the bones of the middle portion of the foot to each other. The Lisfranc ligaments allow for a normal and stable range of motion and shape to the foot.

When the Lisfranc ligaments are disrupted, the stability it had given to the middle of the foot is lost. Attempted activity at the foot will result in pain and abnormal motion. If injury to the Lisfranc ligaments is left untreated, the eventual end result is foot arthritis and deformity.

The current standard orthopaedic treatment of Lisfranc ligament injuries is surgery. The Lisfranc ligaments are fixed by compressing the space between the middle bones of the foot with steel screws. These screws allow for ligament healing. As the ligaments heal, the patient should not resume activity with the fixed foot too soon as the screw may break. A second surgical procedure is often recommended to remove the screw 6 months after surgery. This allows for a complete return of normal foot range of motion, but at the cost of a second procedure.

The use of materials that can be absorbed by the human body to fix the Lisfranc ligaments has only been studied in 1 paper. One such material is the Smart Screw (Bionx, Blue Bell, Pennsylvania) which is approved by the Food and Drug Administration (F.D.A.) and made of polylevolactic acid (PLA). Absorbable screws could be ideal for the treatment of Lisfranc ligament injuries.

Comparing the long-term results of fixing the Lisfranc ligaments with either a steel or absorbable screw is important as there are no studies on the subject to date. There is only 1 published study regarding absorbable screws to fix the Lisfranc ligaments. The purpose of this study is to compare the outcome of steel and absorbable screw fixation of the Lisfranc ligaments in foot injuries in one surgeon's (J.A.) practice at Thomas Jefferson University Hospital, Riddle Memorial Hospital, and Nazareth Hospital.

This study will be conducted in a prospective manner. This study does not focus on experimental procedures or components, but rather involves the accepted management of a select population of patients.

This study will be performed in a randomized, prospective manner involving 2 groups of patients (steel vs. bioabsorbable screw populations) from 3 different hospitals. Power analysis has been conducted to ensure an adequate patient population size.

The risks to patients will be minimal. The standard risks of fixing the Lisfranc ligaments include bleeding, infection, nerve injury, recurrent foot instability, and the dangers of administering anesthesia.

Study Groups Chosen patients for this study will be randomly assigned to one of two groups. Group A will consist of patients that receive the steel screw. Group B will contain the patients that receive the absorbable screw. Postoperative activity restrictions and rehabilitation will be kept the same between the two groups.

Routine protocols for care of foot fracture patients will be utilized regarding infection, wound care, pain control, and weightbearing restrictions. The involved foot will be placed in a non-weight-bearing splint that patients are requested to avoid handling until it is removed by the PI upon the first postoperative visit.

Patients who have their injury fixed using steel screws, need a second surgery in 6 months for removal of the screw. This is the standard textbook treatment and is not a revision surgery. Patients who will receive absorbable screw, wont need this surgery. This will be discussed with the patient at the time of the approach for recruitment.

Outcome evaluation The PI will monitor and follow the patients during and after surgery. Data collection will include the details of the surgery, intraoperative and postoperative course including complications if applicable, and number of revision surgeries performed should they occur. These patients received postoperative follow-up at 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years, and 3 years. Both groups of patients are prohibited from bearing weight on the affected foot for six weeks. Patients will be instructed to gradually increase weight-bearing starting at six weeks.

Postoperative satisfaction and function which will be scored according to the American Orthopaedic Foot and Ankle Society (AOFAS) Midfoot scale which is highly accepted for its validity, reliability, and reproducibility.

Patients will also be asked about their satisfaction with the surgical results using both the 10 cm visual analog scale (VAS) and a four-point scale (poor, mild, good, and excellent). Observed complications including need for further revision surgeries would be documented. All of this information would have been gathered during the patients' follow-up visits in the outpatient clinics after surgery. For those patients that receive a steel screw, they will receive a second outpatient surgical procedure after the 6-month postoperative follow-up to remove that screw using current standard orthopaedic technique.

Postoperative foot X-rays of these patients during their follow up in the outpatient setting will also be examined to view proper alignment and compression of the middle portion of the foot together which indicates healing of the Lisfranc ligaments. Radiographs are used to evaluate the screw for breakage. In the case of the absorbable screw, radiographs are also done to assess absorption.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be adults of any gender or race.
2. Subjects will be adults between 18 and 75 years of age.
3. The underlying diagnosis will be a Lisfranc foot injury.
4. The indication for fixing the Lisfranc ligaments is abnormal separation of the middle part of the foot from each other.
5. Subjects will have received either a steel or absorbable screw to fix the Lisfranc ligaments.

Exclusion Criteria:

1. Subjects may not have any cognitive impairment that would, in the investigator's opinion, preclude study participation or compliance with protocol mandated procedures.
2. Subjects may not have a history of known alcohol, analgesic, or narcotic substance abuse within 12 months prior to pretreatment.
3. Subjects may not have a history of severe psychiatric illness such as depression or psychosis that may influence the results of administered outcome questionnaires.
4. Subjects may not be pregnant.
5. Subjects may be excluded from this study for any reason that may pose unnecessary risk or confounding of data, in the judgment of the investigator. This includes the 4 above points.
6. Subjects must not have intact or normal Lisfranc ligaments in the foot.
7. Subjects may not have a history of deep Lisfranc joint infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measures | 3 years

SECONDARY OUTCOMES:
Visual Analog Score for pain | 3 years
X-rays for maintained healing | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Ahmad, M.D., Principal Investigator — Rothman Institute Orthopaedics
Locations (2):
- United States (2):
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Nazareth Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Thordarson DB, Hurvitz G. PLA screw fixation of Lisfranc injuries. Foot Ankle Int. 2002 Nov;23(11):1003-7. doi: 10.1177/107110070202301106. PMID 12449404